CLINICAL TRIAL: NCT02441426
Title: Etiology, Risk Factors and Interactions of Enteric Infections and Malnutrition and the Consequences for Child Health and Development
Brief Title: Interactions of Enteric Infections and Malnutrition and the Consequences for Child Health and Development
Acronym: MAL-ED
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Foundation for the National Institutes of Health (Other)
Collaborators: University of Virginia (Other); Johns Hopkins University (Other); Aga Khan University (Other); Christian Medical College, Vellore, India (Other); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other); Fogarty International Center of the National Institute of Health (NIH); Penn State University (Other)
Responsible Party: Sponsor
Other Study IDs: MAL-ED-47075
Record Dates: First submitted 2015-05-04; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Diarrhea; Malnutrition; Stunting; Wasting; Immune Response; Cognitive Development
Keywords: Cognitive development; Diarrheal disease; Enteric infections; Malnutrition; Vaccine Response; Enteropathy; Antibiotic use; Micronutrients; Breast feeding; Gut inflammation
MeSH Terms: conditions — Diarrhea; Malnutrition; Growth Disorders; Cachexia; Intestinal Diseases; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, stool, urine, saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Bangladesh: Birth cohort study community in Bangladesh is urban, and located in the Mirpur neighborhood of Dhaka.
  Case control study is being conducted in the same catchment area. Cases defined as children 6-24 months of age with <-2WAZ (weight for age) score, controls are age and community matched with >-1WAZ.
- Brazil: Birth cohort study community in Brazil is urban, and located within the Papoco area of Fortaleza.
  Case control study is being conducted in the same area as the cohort study. Cases are children 6 - 24 months of age, with <-2 WAZ (weight for age) score, controls are age and community matched children with >-1 WAZ.
- India: Birth cohort study community in India is urban, and located in the southern state of Tamil Nadu, specifically in Vellore.
- Nepal: Birth cohort study community in Nepal is semi-urban, and located in Bhaktapur, approximately 25km from Kathmandu.
- Pakistan: Birth cohort study community in Pakistan is rural, and located in Naushero Feroze, Sindh.
- Peru: Birth cohort study community in Peru is rural, and located approximately 15km from Iquitos in Loreto.
- South Africa: Birth cohort study community in South Africa is rural/peri-urban, and comprised of nine settlements within Limpopo Province.
- Tanzania: Birth cohort study community in Tanzania is rural, and located within Haydom.

SUMMARY:
Malnutrition is considered one of the most prevalent risk factors for morbidity and mortality in children under five. An estimated 20% of children in the developing world are malnourished [1] and poor nutrition is linked to more than half of all child deaths worldwide [2]. Malnutrition in early childhood may lead to cognitive and physical deficits and may cause similar deficits in future generations as malnourished mothers give birth to low birth weight children [3]. In addition, malnutrition increases susceptibility and incidence of infections and is associated with diminished response to vaccines.

The MAL-ED Project is designed to determine the impact of enteric infections/diarrhea that alter gut function and impair children's nutrition, growth and development to help develop new intervention strategies that can break the vicious enteric infection-malnutrition cycle and reduce its global burden.

The overall objective of the MAL-ED Project is to quantify the associations of specific enteric pathogens, measures of physical and mental development, micronutrient malnutrition, gut function biomarkers, the gut microbiome, and immune responses in very young children in resource-limited settings across eight sites that vary by culture, economics, geography, and climate.

The central hypothesis of the MAL-ED Project is that infection (and co-infection) with specific enteropathogens leads to impaired growth and development and to diminished immune response to orally administered vaccines by causing intestinal inflammation and/or by altering intestinal barrier and absorptive function. Data analyses will test for associations between enteropathogen infections and growth/development to help illuminate:

* which micro-organisms or mixed infections are most frequently associated with growth faltering and poor development; and
* at what age specific infections cause the most disruption to growth and development and impair immune response.

ELIGIBILITY:
Inclusion Criteria:

* Less than 17 days old.

Exclusion Criteria:

* Mother is less than 16 years of age.
* Mother has another child inthe MAL-ED study.
* Pregnancy resulted in multiple birth (e.g., twins).
* Child has a severe disease requiring hospitalization for something other than for a typical healthy birth.
* Child has a severe or chronic condition diagnosed by a medical doctor (e.g., neonatal disease, renal disease, chronic heart failure, liver disease, cystic fibrosis, congenital conditions).
* Child has enteropathies diagnosed by medical doctor.
* Mother is living and unable to provide informed consent.

Ages: 1 Minute to 17 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population for the MAL-ED Project is a birth cohort. Pregnant women were identified from their communities, consented and the child will be enrolled.
Sampling Method: Probability Sample
Enrollment: 1796 (Estimated)
Dates: Start 2008-11; Primary Completion 2017-02 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Diarrhea | Each diarrheal episode willbe recorded for up to 24 months of age.
  All diarrheal samples are analyzed for the presence of bacterial, viral, and parasitic pathogens. Normal stool is collected monthly and analyzed for the same list of 57 different pathogens.
Anthropometry | Anthropomentry will be recorded each month for up to 24 months of age.
  Head Circumference, length, and weight are measured monthly on the anniversary of the child's birth.
Cognitive development | Cognitive development will be recorded at 6 months of age.
  A battery of tests include the Bayley Scales of Infant Development, MacArthur Words and Gestures, Infant Temperament Scale, HOME inventory, SRQ-20 and Raven's Combined Progressive Matrices.
Vaccine response | Vaccine response will be recorded at 7 months of age.
  Antibody titers will be determined following immunization against rotavirus, polio virus, tetanus toxoid, pertussis toxin and measles vaccines.
Cognitive development | Cognitive development will be recorded at 8 months of age.
  A battery of tests include the Bayley Scales of Infant Development, MacArthur Words and Gestures, Infant Temperament Scale, HOME inventory, SRQ-20 and Raven's Combined Progressive Matrices.
Cognitive development | Cognitive development will be recorded at 15 months of age.
  A battery of tests include the Bayley Scales of Infant Development, MacArthur Words and Gestures, Infant Temperament Scale, HOME inventory, SRQ-20 and Raven's Combined Progressive Matrices.
Vaccine response | Vaccine response will be recorded at 15 months of age.
  Antibody titers will be determined following immunization against rotavirus, polio virus, tetanus toxoid, pertussis toxin and measles vaccines.
Cognitive development | Cognitive development will be recorded 24 months of age.
  A battery of tests include the Bayley Scales of Infant Development, MacArthur Words and Gestures, Infant Temperament Scale, HOME inventory, SRQ-20 and Raven's Combined Progressive Matrices.
Vaccine response | Vaccine response will be recorded at 24 months of age.
  Antibody titers will be determined following immunization against rotavirus, polio virus, tetanus toxoid, pertussis toxin and measles vaccines.

SECONDARY OUTCOMES:
Gut inflammation | Gut inflammation will be recorded each month for up to 24 months of age.
  Stool biomarkers will be evaluated to detect gut and systemic inflammation.
Gut integrity | Gut integritywill be recorded at at 3 months of age.
  Intestinal absorptive capacity and barrier function will be assessed by dual sugar permeability test.
Gut integrity | Gut integritywill be recorded at at 6 months of age.
  Intestinal absorptive capacity and barrier function will be assessed by dual sugar permeability test.
Gut integrity | Gut integritywill be recorded at at 9 months of age.
  Intestinal absorptive capacity and barrier function will be assessed by dual sugar permeability test.
Gut integrity | Gut integritywill be recorded at at 15 months of age.
  Intestinal absorptive capacity and barrier function will be assessed by dual sugar permeability test.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gottlieb, Ph.D., Principal Investigator — Fountation for the National Institutes of Health; Roger Glass, M.D., Principal Investigator — Fogarty International Center of the National Institute of Health
Locations (8):
- International Centre for Diarrheal Disease Research, Bangladesh, Dhaka, Bangladesh
- Universidade Federal do Ceará, Fortaleza, Brazil
- Christian Medical College, Vellore, India
- Institute of Medicine, Kathmandu, Nepal
- Aga Khan University, Karachi, Pakistan
- JHSPH Satellite Laboratory, Iquitos, Peru
- University of Venda, Limpopo, South Africa
- Haydom Lutheran Hospital, Haydom, Tanzania

REFERENCES:
- [Derived] Nemati K, Michael YZ, Hhando BP, Jatosh S, Houpt ER, Mduma E, DeBoer MD. Catch-up growth following early-life stunting in a low-resource area in rural Tanzania: the MAL-ED Metabolic study. BMJ Open. 2025 Aug 21;15(8):e100955. doi: 10.1136/bmjopen-2025-100955. PMID 40840991
- [Derived] Arndt MB, Richardson BA, Mahfuz M, Ahmed T, Haque R, Gazi MA, John-Stewart GC, Denno DM, Scarlett JM, Walson JL; coordination with The Interactions of Malnutrition & Enteric Infections: Consequences for Child Health and Development Project Network. Plasma Fibroblast Growth Factor 21 Is Associated with Subsequent Growth in a Cohort of Underweight Children in Bangladesh. Curr Dev Nutr. 2019 Mar 30;3(5):nzz024. doi: 10.1093/cdn/nzz024. eCollection 2019 May. PMID 31093598
- [Derived] Colston JM, Ahmed T, Mahopo C, Kang G, Kosek M, de Sousa Junior F, Shrestha PS, Svensen E, Turab A, Zaitchik B; MAL-ED Network. Evaluating meteorological data from weather stations, and from satellites and global models for a multi-site epidemiological study. Environ Res. 2018 Aug;165:91-109. doi: 10.1016/j.envres.2018.02.027. Epub 2018 Apr 21. PMID 29684739
- [Derived] Colston JM, Penataro Yori P, Colantuoni E, Moulton LH, Ambikapathi R, Lee G, Rengifo Trigoso D, Siguas Salas M, Kosek MN. A methodologic framework for modeling and assessing biomarkers of environmental enteropathy as predictors of growth in infants: an example from a Peruvian birth cohort. Am J Clin Nutr. 2017 Jul;106(1):245-255. doi: 10.3945/ajcn.116.151886. Epub 2017 Jun 7. PMID 28592604
- [Derived] Platts-Mills JA, Taniuchi M, Uddin MJ, Sobuz SU, Mahfuz M, Gaffar SA, Mondal D, Hossain MI, Islam MM, Ahmed AS, Petri WA, Haque R, Houpt ER, Ahmed T. Association between enteropathogens and malnutrition in children aged 6-23 mo in Bangladesh: a case-control study. Am J Clin Nutr. 2017 May;105(5):1132-1138. doi: 10.3945/ajcn.116.138800. Epub 2017 Apr 5. PMID 28381477